CLINICAL TRIAL: NCT07092943
Title: A Comparison of Driving Pressure Guided Mechanical Ventilation With Lung Protective Ventilation Among Patients Presenting for Elective Surgeries at a Tertiary Care Hospital; A Randomized Control Trial
Brief Title: Driving Pressure Guided Mechanical Ventilation Versus Lung Protective Ventilation Among Patients Undergoing Elective Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Huda Tariq, Principal Investigator, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 200/IREF/RMU/2025
Record Dates: First submitted 2025-07-20; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mechanical Ventilation; Lung Protective Ventilation; Driving Pressure
Keywords: General Anesthesia; Mechanical ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lung Protective ventilation (Sham Comparator)
  Interventions: Device: Lung protective ventilation
- Driving pressure guided ventilation (Experimental)
  Interventions: Device: Driving pressure guided ventilation

INTERVENTIONS:
Device: Lung protective ventilation — The patient in this group will receive tidal volume at 6-8 ml/kg of ideal body weight with PEEP of 5 cm of H2O and plateau pressure will be kept less than 30cm of H2O.
  Arms: Lung Protective ventilation
Device: Driving pressure guided ventilation — They will receive tidal volume of 6-8 ml/kg of ideal body weight and initial PEEP of 5 cm of water. Principal investigator will then incrementally increase PEEP by 2 cm of water till a value 15 cm of water PEEP is reached or Plateau pressure becomes equal to 30 cm of water or driving pressure starts to increase or there is change in any hemodynamics. Each incremental PEEP will last for 3 respiratory cycles before moving on to next value. PEEP value with lowest driving pressure will then be selected for the duration of surgical procedure
  Arms: Driving pressure guided ventilation

SUMMARY:
Patient undergoing surgeries in general anesthesia require support of their breathing by ventilator. Different strategies can be used to manage breathing of the patient. Lung protective ventilation provides breathing at a set volume determined by patient ideal body weight, along with a set rate to maintain adequate breathing. The pressures in the lower airway are kept less than 30 cm of H20 while a pressure of 5cm of H20 is applied to prevent lung collapse. Recently to above mentioned regimen a driving pressure is added which is a difference between lower airway pressure and pressure applied to prevent lung collapse. Ventilatory settings are adjusted to keep this driving pressure less than 15 cm of H2O.

DETAILED DESCRIPTION:
Lung protective ventilation provides tidal volume at 6-8 ml/kg along with a set respiratory while keeping plateau pressure less than 30cm of H2O and Peak pressure less than 35cm of H2O and PEEP of 5cm of H20 is applied. The aim is to prevent volutrauma, barotrauma and atelectrauma. To above mentioned regimen another parameter is added that is driving pressure. It is manipulated by adjusting PEEP level so that difference between Plateau Pressure and PEEP is less than equal to 15cm of water.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class: I and II.
* Elective laparoscopic surgeries requiring General Anesthesia and Mechanical ventilation
* Patients receiving neuromuscular blockade during surgery.
* Receiving Mechanical ventilation for at least 1h.

Exclusion Criteria:

* Pregnancy
* Patients who had received mechanical ventilation of more than 1h in the previous 2 weeks.
* Body mass index >35 kg/m2
* Smokers and ASA class III and above.
* Thoracic and Cardiac surgery

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Intra-operative pulmonary compliance | This will be measured at 10 minutes interval in the intraoperative period and then mean will be calculated.

SECONDARY OUTCOMES:
Oxygenation index | This will be the ratio of PaO2/FiO2 and this will be measured during surgery (at time of skin closure)
PEtCO2-PaCO2 gradient | This will be the PEtCO2-PaCO2 gradient and this will be measured during surgery (at time of skin closure)
Intra-operative blood pressure | This will be Systolic, Diastolic and Mean Blood pressure measured at baseline and then 10 minutes interval in the intraoperative period. Mean will be calculated for comparison across groupss.
Post operative pulmonary complications | This will be the need for prolonged ventilatory support, need for re-intubation ,need for supplemental oxygenation and its duration, PaO2/FiO2 ratio less than 300, pneumothroax. These will be observed in first 24hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park M, Yoon S, Nam JS, Ahn HJ, Kim H, Kim HJ, Choi H, Kim HK, Blank RS, Yun SC, Lee DK, Yang M, Kim JA, Song I, Kim BR, Bahk JH, Kim J, Lee S, Choi IC, Oh YJ, Hwang W, Lim BG, Heo BY. Driving pressure-guided ventilation and postoperative pulmonary complications in thoracic surgery: a multicentre randomised clinical trial. Br J Anaesth. 2023 Jan;130(1):e106-e118. doi: 10.1016/j.bja.2022.06.037. Epub 2022 Aug 20. PMID 35995638
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35995638/